CLINICAL TRIAL: NCT04453618
Title: Safety, Tolerability, Pharmacokinetics, and Food Effect of a Tablet Formulation of SYHA1402 in Healthy Subjects: A Phase-1, Single Center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Food Effect of SYHA1402 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HA1403-CSP-002；V1.0
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Peripheral Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Food effect (Experimental): Healthy subjects receive a single dose of SYHA1402 (100mg) in either a fasted state or with a meal.
  Interventions: Drug: FE-SYHA1402 100mg
- Multiple doses 25mg (Experimental): Healthy subjects receive multiple doses of SYHA1402 (25mg) or Placebo(25mg) for a total of 7 days (QD on Day1 and Day7, Q8h on Day2 to Day6）.
  Interventions: Drug: SYHA1402-25mg; Drug: Placebo-25mg
- Multiple doses 50mg (Experimental): Healthy subjects receive multiple doses of SYHA1402 (50mg) or Placebo (50mg) for a total of 7 days (QD on Day1 and Day7, Q8h on Day2 to Day6）.
  Interventions: Drug: SYHA1402-50mg; Drug: Placebo-50mg
- Multiple doses 150mg (Experimental): Healthy subjects receive multiple doses of SYHA1402 (150mg) or Placebo (150mg) for a total of 7 days (QD on Day1 and Day7, Q8h on Day2 to Day6）.
  Interventions: Drug: SYHA1402-150mg; Drug: Placebo-150mg

INTERVENTIONS:
Drug: FE-SYHA1402 100mg — in either a fasted state or with a meal
  Arms: Food effect
Drug: SYHA1402-25mg — SYHA1402 25mg, oral tablets
  Arms: Multiple doses 25mg
Drug: Placebo-25mg — Matching placebo tablets
  Arms: Multiple doses 25mg
Drug: SYHA1402-50mg — SYHA1402 50mg, oral tablets
  Arms: Multiple doses 50mg
Drug: Placebo-50mg — Matching placebo tablets
  Arms: Multiple doses 50mg
Drug: SYHA1402-150mg — SYHA1402 150mg, oral tablets
  Arms: Multiple doses 150mg
Drug: Placebo-150mg — Matching placebo tablets
  Arms: Multiple doses 150mg

SUMMARY:
A Multiple Doses Study to Evaluate the Safety, Tolerability, Pharmacokinetics (Including Food Effect) of SYHA1402 in Healthy Subjects.

DETAILED DESCRIPTION:
This study consists of two parts: The objective of the food effect study (Part 1) is to investigate the effect of food on the pharmacokinetic profiles of SYHA1402 tablets under fed and fasted conditions following the oral administration of SYHA1402.

The primary objective of the multiple doses study (Part 2) is to investigate safety, tolerability and Pharmacokinetics of SYHA1402 in healthy subjects following oral administration of Multiple rising doses.

Secondary objectives are the exploration of pharmacokinetics (PK) following multiple oral doses.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18 to 45 years (inclusive).
2. Have a body mass index (BMI) between 19.0 and 26.0 kg/m2 inclusive and weigh at least 45.0 kg (female) or 50.0 kg (male) inclusive at screening.
3. With no clinically significant or relevant abnormalities as determined by medical history, vital signs, physical examination, and clinical laboratory tests.
4. All subjects of reproductive potential must agree to use effective, non-hormonal contraceptive measures (such as condoms, intrauterine devices without drugs) from the signing of informed consent to 3 months after the study. A subject is eligible to participate if she/he is not a person of childbearing potential (had a bilateral oophorectomy, bilateral salpingo-oophorectomy, or vasectomy). A male subject refrains from donating sperm during the study period and for 3 months after the study.
5. Signed informed consent form.

Exclusion Criteria:

1. Female subjects who are pregnant or lactating.
2. History or current evidence of any clinically significant cardiac, endocrinologic, hematologic, hepatobiliary, immunologic, metabolic, urologic, pulmonary, neurologic, psychiatric, renal, or other major disease, as determined by the investigator.
3. Surgery history within six months before signing the informed consent;
4. Allergic history to more than one drug or other serious allergic history.
5. Any other abnormal findings on vital signs
6. Any clinically significant abnormalities in ECG: a QTc interval greater than 450 ms (male) or 470 ms (female), or with a history of prolonged QTc interval;
7. Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (anti-HCV), Human immunodeficiency virus antibody (anti-HIV) or Treponema Pallidum antibody (Anti-TP) at screening.
8. Use of drugs within 2 weeks before signing the informed consent, including over-the-counter or prescription medication, including biological product, Chinese traditional medicine, herbal medicine, vitamin dietary supplements, health care products, oral or imbedded long-acting contraceptives.
9. Alcohol abuse or positive test for alcohol screening.
10. Smoker.
11. History or clinical evidence of drug abuse within the one years before screening, or positive test for drug abuse at screening.
12. Use of too much caffeine in beverages, foods or in any form, which may interfere the absorption, distribution, metabolism, or excretion of drugs, within 4 weeks before signing informed consent
13. Loss of blood or blood donation more than 200 mL within 8 weeks before signing informed consent, or plan on blood donation during the study period and 1 months after the last dose of drug.
14. Have a surgical schedule or a plan on excessive physical activity during the study period.
15. Subjects participating in other clinical trials, or who have participated in any other clinical trials of drugs within three months before signing informed consent;
16. Not suitable for this trial as determined by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Effect of food on the pharmacokinetic(Cmax） | Predose and multiple timepoints up to 24 hours after the last dose in fed and fasted conditions
  Effect of food on the pharmacokinetic profile of SYHA1402 based on maximum observed plasma concentration (Cmax) (Part 1).
Effect of food on the pharmacokinetic(AUC0-inf） | Predose and multiple timepoints up to 24 hours after the last dose in fed and fasted conditions
  Effect of food on the pharmacokinetic profile of SYHA1402 based on AUC0-inf (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to infinity) (Part 1).
Effect of food on the pharmacokinetic(AUC0-t） | Predose and multiple timepoints up to 24 hours after the last dose in fed and fasted conditions
  Effect of food on the pharmacokinetic profile of SYHA1402 based on AUC0-t (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to time of last measurable concentration) (Part 1).
Safety and tolerability of multiple doses of SYHA1402 administered orally will be assessed (Part2). | up to 5 days after the last dose
  incidence and severity of adverse events (AEs), abnormalities in clinical laboratory assessments, ECGs, vital sign assessments, and physical exams

SECONDARY OUTCOMES:
Safety and tolerability of SYHA1402 administered orally in fed and fasted conditions will be assessed (Part1) | up to 4 days after the last dose
  incidence and severity of adverse events (AEs), abnormalities in clinical laboratory assessments, ECGs, vital sign assessments, and physical exams
AUC0-t(Part2) | Predose and multiple timepoints up to 24 hours after the last dose
  Rate and Extent of Absorption SYHA1402 by Assessment of the area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point
AUC0-inf(Part2) | Predose and multiple timepoints up to 24 hours after the last dose
  Rate and Extent of Absorption SYHA1402 by Assessment of the area under the concentration-time curve of the analyte in plasma over the time interval from 0 to infinity
Cmax(Part2) | Predose and multiple timepoints up to 24 hours after the last dose
  Rate and Extent of Absorption SYHA1402 by Assessment of the maximum measured concentration of the analyte in plasma
Tmax(Part2) | Predose and multiple timepoints up to 24 hours after the last dose
  Rate and Extent of Absorption SYHA1402 by Assessment of the Time to Reach Maximum Observed Concentration
t1/2z(Part2) | Predose and multiple timepoints up to 24 hours after the last dose
  Rate and Extent of Absorption SYHA1402 by Assessment of the Apparent Terminal Elimination Half-life
CL/F(Part2) | Predose and multiple timepoints up to 24 hours after the last dose
  Rate and Extent of Absorption SYHA1402 by Assessment of the Apparent Clearance
Vz/F(Part2) | Predose and multiple timepoints up to 24 hours after the last dose
  Rate and Extent of Absorption SYHA1402 by Assessment of the Apparent Volume of Distribution
Rac(AUC)(Part2) | Predose and multiple timepoints up to 24 hours after the last dose
  Rate and Extent of Absorption of SYHA1402 by Assessment of the Accumulation Ratio
Rac(Cmax) (Part2) | Predose and multiple timepoints up to 24 hours after the last dose
  Rate and Extent of Absorption of AZD7986 by Assessment of the Accumulation Ratio for Cmax
The assessment of the dose-proportionality based on Cmax (Part2) | Predose and multiple timepoints up to 24 hours after the last dose
  The assessment of the dose-proportionality in the plasma pharmacokinetics (Cmax) of SYHA1402
The assessment of the dose-proportionality based on AUC (Part2) | Predose and multiple timepoints up to 24 hours after the last dose
  The assessment of the dose-proportionality in the plasma pharmacokinetics (AUC) of SYHA1402